CLINICAL TRIAL: NCT02235025
Title: Ventilatory Constraints During Exercise in Asymptomatic Versus Symptomatic Patients With Mild COPD
Brief Title: Asymptomatic Versus Symptomatic Mild COPD: Comparisons at Rest and at Exercise
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Besancon (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: BAL-1
Record Dates: First submitted 2014-08-27; First posted 2014-09-09 (Estimated); Last update posted 2014-09-09 (Estimated); Status verified 2014-08

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: mild COPD; dyspnea; exercise; respiratory mechanics
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Dyspnea; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Asymptomatic mild COPD (Other): Subjects of this group have GOLD grade I COPD (post-bronchodilator FEV1 > 80% predicted and FEV1/FVC < 0.7). They also have a modified Medical Research Council (mMRC) score equal to zero and are free of respiratory symptoms including chronic cough and/or chronic expectoration and/or chronic wheeze.
  Interventions: Other: Cardio-pulmonary exercise testing
- Symptomatic mild COPD (Other): Subjects of this group have GOLD grade I COPD (post-bronchodilator FEV1 > 80% predicted and FEV1/FVC < 0.7). They also have a modified Medical Research Council (mMRC) score > 0.
  Interventions: Other: Cardio-pulmonary exercise testing
- Healthy controls (Other): Healthy controls have normal baseline spirometry (FEV1 > 80% predicted, FEV1/FVC > 0.7). They don't have any health problems, including cardiovascular, metabolic, neuromuscular, musculoskeletal, or respiratory diseases that could contribute to breathlessness or exercise limitation. They have a mMRC score equal to zero and do not complain any respiratory symptoms including chronic cough and/or chronic expectoration and/or chronic wheeze and/or chronic respiratory related medication.
  Interventions: Other: Cardio-pulmonary exercise testing

INTERVENTIONS:
Other: Cardio-pulmonary exercise testing

SUMMARY:
The current definition of chronic obstructive pulmonary disease (COPD) is based on the presence of persistent airflow obstruction assessed by spirometry. About half of the subjects with mild COPD (i.e. reduced forced expiratory volume in one second (FEV1) on forced vital capacity (FVC) ratio along with normal FEV1] are asymptomatic. Subjects with symptomatic mild COPD have reduced exercise tolerance and abnormal dynamic ventilatory mechanics compared to healthy subjects. The physiological and perceptual responses to exercise of subjects with asymptomatic mild COPD are currently unknown.

The purpose of this study is to assess exercise tolerance, ventilatory constraints on tidal volume expansion and dyspnoea in asymptomatic mild COPD subjects undergoing incremental cycle cardiopulmonary exercise testing (CPET) to the limit of tolerance compared with symptomatic mild COPD and healthy controls.

DETAILED DESCRIPTION:
Subjects attend one single visit. If needed, COPD subjects are asked to stop any respiratory related medication such as short and long acting bronchodilators 72 hours prior to the visit. Subjects are asked to arrive early in the morning. After informed consent and appropriate screening of medical history, all subjects complete the mMRC scale. A complete medical history is collected. Subjects thereafter complete pulmonary function testing pre- and 30-min post-bronchodilator. Subjects are given a normal mixed meal and are asked not to drink alcohol or coffee.

A symptom-limited incremental cycle exercise test is performed on the same day, at least 6 hours after the bronchodilator test and at least 4 hours after the meal. After a steady-state resting period, a 3-min warm-up is conducted at about 20% of individually estimated maximal work load (Wmax), and the load is increased every minute in such a way that the test duration is >8 and <12 min. The following data are obtained breath by breath and expressed as 30-s averages: V'O2 and carbon dioxide production (V'CO2); minute ventilation (V'E); tidal volume (VT); respiratory rate; and ventilatory equivalents for oxygen and carbon dioxide. Blood pressure is measured every minute by a sphygmomanometer. Blood samples are withdrawn from the arterialized earlobe at rest and at near-maximal exercise. Tests are terminated at the point of symptom limitation (peak exercise). Upon exercise cessation, subjects are asked to verbalize their main reason for stopping exercise (breathing discomfort, leg discomfort or both).

ELIGIBILITY:
Inclusion Criteria:

* For COPD groups: post-bronchodilator forced expiratory volume in 1 sec (FEV1) ≥ 80% predicted and a FEV1/forced vital capacity (FVC) ratio < 0.70
* For the "Asymptomatic mild COPD" group: modified Medical Research Council (mMRC) score equal to zero and absence of respiratory symptoms including chronic cough and/or chronic expectoration and/or chronic wheeze.
* For the "Symptomatic mild COPD" group: mMRC) score > 0
* For the "Healthy controls" group: FEV1 > 80% predicted and FEV1/FVC > 0.7) and a mMRC score equal to zero and absence of respiratory symptoms including chronic cough and/or chronic expectoration and/or chronic wheeze
* Able to perform all study procedures and provide informed consent

Exclusion Criteria:

* Presence of a medical condition other than COPD that could cause or contribute to breathlessness (i.e., a respiratory disease other than COPD and/or a metabolic and/or a cardiovascular disease)
* Presence of disorders other than COPD that could interfere with exercise testing, such as neuromuscular diseases or musculoskeletal problems
* History or clinical evidence of asthma
* Use of daytime oxygen or exercise-induced arterial oxygen desaturation to <80% on room air

Min Age: 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 111 (Actual)
Dates: Start 2012-09; Primary Completion 2013-08 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
Dyspnea intensity measured by the 10-point Borg scale during cycle exercise | up to 12 minutes
  Dyspnea intensity is measured at rest and every two minutes thereafter. Dyspnea intensity at 80% of maximal predicted work rate is calculated by linear interpolation between adjacent measurement points for each subject

SECONDARY OUTCOMES:
Inspiratory capacity | up to 12 minutes
  Inspiratory capacity as a function of work rate is studied as a continuous variable. In addition, a decrease in inspiratory capacity from rest of more than 150 mL at any time-point during exercise defines dynamic hyperinflation
Tidal volume as a function of minute ventilation | up to 12 minutes
  In the relationship between tidal volume (VT) and minute ventilation (V'E), there is an inflection point beyond which almost no further change in VT is possible despite a continued increase in V'E. This inflection in the VT response marks the point were dyspnoea sharply raises because of mechanical constraints on VT expansion. This inflection point is determined for each patient by analyzing individual Hey plot

CONTACTS AND LOCATIONS:
Overall Officials: Bruno Degano, MD, PhD, Principal Investigator — CHU Besançon, France
Locations (1):
- Department of respiratory diseases, Besançon, France